CLINICAL TRIAL: NCT07072312
Title: Feasibility, Acceptability and Fidelty of Integrating Navigation to Improve Adherence: Tobacco Treatment Program for Cancer Patients A Pragmatic Pilot Study
Brief Title: Feasibility, Acceptability and Fidelity of Integrating a Navigation Intervention Into Tobacco Treatment Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Temple University (Other)
Responsible Party: Principal Investigator, Linda Fleisher, Research Professor, Fox Chase Cancer Center
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-1011
Record Dates: First submitted 2024-03-01; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Cancer
Keywords: Tobacco Cessation; Patient Navigation
MeSH Terms: conditions — Neoplasms; Tobacco Use Cessation

STUDY DESIGN:
Intervention Model Description: The first 30 patients are enrolled to the pre-intervention group and receive standard of care to serve as a comparison group. The subsequent patients are enrolled to the single arm to receive the standard care and patient navigation intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient Navigation (Experimental): Participants receive patient navigation after their first and second tobacco treatment visits.
  Interventions: Behavioral: Adjuvant Patient Navigation for Tobacco Treatment

INTERVENTIONS:
Behavioral: Adjuvant Patient Navigation for Tobacco Treatment — Patients in the study meet with the Patient Navigator two weeks after their first tobacco treatment visit and again after their second visit with the Tobacco Treatment Provider. The Patient Navigator will discuss psychosocial and other cessation barriers. The Patient Navigator will connect the patients with appropriate resources to help overcome these barriers.

SUMMARY:
Patient Navigation is being included as part of a tobacco treatment program for cancer patients to help patients overcome barriers to quitting.

DETAILED DESCRIPTION:
The primary objective of this prospective, interventional pilot study is to assess the feasibility, acceptability and fidelity of a navigation intervention embedded into the clinical Tobacco Treatment Program.

The investigators will employ a pre-post design with two cohorts (30 to the pre-intervention, and 90 to the intervention, respectively) to address the specific aims of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a cancer diagnosis. Patients may be undergoing active therapy or may have completed treatment.
2. English speaking.
3. Age > 18 years.
4. Active tobacco cigarette user, defined as having smoked a cigarette within the 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Feasibility of Integrating Navigation into Tobacco Treatment Program | Prior to first TTP visit - consented and enrolled
  The number of patients who enroll and consent to receiving the tobacco treatment program navigation intervention. Feasibility will be obtained if at least 60% consent and enroll.
Patient Acceptability of Navigation in Tobacco Treatment - Patient Recommendation | One and six months post initial navigation intervention
  The number of patients who state they would likely or highly likely to recommend the service to other cancer patients. Acceptability will obtained if 70% of patients likely recommend the service.
Provider Implementation of the Intervention -Fidelity to Protocol | Baseline to 6 months
  The number of patients who receive the two primary components of the navigation intervention, assessing tobacco cessation barriers and psychosocial barriers. Fidelity will be achieved if 80% of cases include both elements measured through a review of the navigation case management system.
Fidelity of Utilization of Navigation Intervention - Patient Participation | Baseline to 6 months
  Number of patients who had at least 2 navigation encounters. Fidelity will be achieved if 80% of patients have a minimum of 2 navigation encounters through the navigation case management review.

SECONDARY OUTCOMES:
7-Day Point Prevalence | Six months
  7-Day point prevalence of tobacco will be assessed at six month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Fleisher, PhD, MPH, Principal Investigator — Temple Univeristy Health System - Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No